CLINICAL TRIAL: NCT04515888
Title: Evaluation of the Prevalence of Pelvic Static Disorders in Women Treated for Localized Breast Cancer During Adjuvant Hormone Therapy.
Brief Title: Evaluation of the Prevalence of Pelvic Static Disorders in Women With Localized Breast Cancer
Acronym: STATICBREAST
Status: Completed | Type: Observational
Sponsor: Institut du Cancer de Montpellier - Val d'Aurelle (Other)
Responsible Party: Sponsor
Other Study IDs: PROICM 2020-01 OST
Record Dates: First submitted 2020-08-07; First posted 2020-08-17 (Actual); Last update posted 2021-11-04 (Actual); Status verified 2021-11

CONDITIONS: Breast Cancer
Keywords: localized breast cancer; pelvic static disorders; hormontherapy
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- target population: The target population of the study consists of breast cancer female patients over 50 years old followed for an invasive carcinoma expressing hormone receptors, non metastatic, undergoing adjuvant hormone therapy.
  Interventions: Other: PFDI-20 / PFIQ-7 questionnaires
- control population: The control group will be composed of patients followed for an in situ carcinoma treated by surgery +/- radiotherapy, without hormone therapy.
  Interventions: Other: PFDI-20 / PFIQ-7 questionnaires

INTERVENTIONS:
Other: PFDI-20 / PFIQ-7 questionnaires — PFDI-20 / PFIQ-7 questionnaires (one shot)

SUMMARY:
In this study, investigator propose to assess the prevalence of pelvic static disorders in women undergoing adjuvant hormone therapy for localized breast cancer and to assess the overall quality of life in these patients

DETAILED DESCRIPTION:
Breast cancer is the most common cancer in women. Its incidence increases with 58,459 new cases in France in 2018, however its mortality decreases with a survival rate of 87% at 5 years.

Therapeutic options are surgery, radiotherapy, chemotherapy and hormone therapy. Hormone therapy is one of the major treatments for hormone-sensitive tumors with a prescription made in around 70% of breast cancer cases. These different hormone therapies cause a hormonal imbalance with in particular an important anti-estrogenic action. Hormonal deprivation and menopause can be responsible for the occurrence of pelvic statics disorder.[5-9] Pelvic static disorder (PTS) is a common problem for women, which can occur at any age.

These disorders include urinary incontinence, stress or urgency, anal incontinence, genital prolapse.

Hypothesis's investigator is that hormone therapy may be responsible for PTS. In this study, investigator propose to assess the prevalence of pelvic static disorders in women undergoing adjuvant hormone therapy for localized breast cancer and to assess the overall quality of life in these patients.

ELIGIBILITY:
Inclusion Criteria:

* Women with Age ≥ 50 years
* Menopaused
* Patient followed for carcinoma in situ or infiltrating the breast with or without hormone therapy
* Patient who was treated by surgery after June 2015, whether or not followed by radiotherapy or chemotherapy.
* Patient who agreed, after receiving information, to participate to the study.

Exclusion Criteria:

* Metastatic breast cancer
* Patient with a history of pelvic static surgery
* Patient with a history of pelvic irradiation
* Patient unable or unwilling to complete the questionnaires
* Patient with a history of urinary incontinence treatment
* Patient not affiliated to the French social security system
* Subject under tutelage, curatorship or safeguard of justice,
* Patient in an emergency situation,
* Patient whose regular monitoring is impossible for psychological, family, social or geographical reasons,
* Pregnant and / or breastfeeding woman.

Min Age: 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The target population of the study consists of breast cancer female patients over 50 years old followed for an invasive carcinoma expressing hormone receptors, non metastatic, undergoing adjuvant hormone therapy. The control group will be composed of patients followed for an in situ carcinoma treated by surgery +/- radiotherapy, without hormone therapy
Sampling Method: Probability Sample
Enrollment: 246 (Actual)
Dates: Start 2020-09-18 (Actual); Primary Completion 2021-02-12 (Actual); Study Completion 2021-07-06 (Actual)

PRIMARY OUTCOMES:
Evaluate the prevalence of pelvic static disorders in patients treated for localized breast cancer and undergoing adjuvant hormone therapy (Hormontherapy +). | Day 1
  Pelvic static disorders rate according to the Questionnaire on pelvic static disorders PFDI-20 in patients (hormonotherapy +)

SECONDARY OUTCOMES:
Evaluate the prevalence of pelvic static disorders in patients (hormonotherapy -) | Day 1
  Pelvic static disorders rate according to the Questionnaire on pelvic static disorders PFDI-20 in patients hormonotherapy -
Compare the prevalence of Pelvic static disorders between the 2 groups Hormonotherapy - /Hormonotherapy + | Day 1
  Pelvic static disorders rate according to the Questionnaire on pelvic static disorders PFDI-20 in patients hormonotherapy - and patient hormontherapy +
Evaluate the impact of pelvic static disorders on quality of life | Day 1
  Estimation of quality of life according to the PFIQ-7 (Pelvic Floor Impact Questionnaire) in the 2 populations. the total score of the PFIQ-7 is obtained by adding the scores for each scale (between 0 (no impact) and 300 (maximum impact))
Estimate pelvic symptoms in the hormone therapy (Hormonotherapy +) / Non hormone therapy (Hormonotherapy -) groups | Day 1
  Estimation of pelvic symptoms scores according to the PFDI-20 (Pelvic Floor Distress Inventory) questionnaire in the 2 populations. the total score of the PFDI-20 is obtained by adding the scores for each scale (between 0 (no impact) and 300 (maximum impact))
Evaluate the correlation between hormone therapy and pelvic static disorders | Day 1
  Estimate the Rational rate between pelvic static disorders and hormone therapy with adjustment on known parameters : age, obesity, type of birth (vaginal or caesarean)
Research the risk factors for pelvic static disorders | Day 1
  number of risk factors based on data collected

CONTACTS AND LOCATIONS:
Overall Officials: Laure DELMOND, MD, Study Chair — ICM Val d'Aurelle
Locations (1):
- Icm Val D'Aurelle, Montpellier, Herault, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Cowppli-Bony A, Colonna M, Ligier K, Jooste V, Defossez G, Monnereau A; le Reseau Francim; Reseau des registres de cancer Francim. [Descriptive epidemiology of cancer in metropolitan France: Incidence, survival and prevalence]. Bull Cancer. 2019 Jul-Aug;106(7-8):617-634. doi: 10.1016/j.bulcan.2018.11.016. Epub 2019 Mar 2. French. PMID 30833045
- [Result] Jones SE, Cantrell J, Vukelja S, Pippen J, O'Shaughnessy J, Blum JL, Brooks R, Hartung NL, Negron AG, Richards DA, Rivera R, Holmes FA, Chittoor S, Whittaker TL, Bordelon JH, Ketchel SJ, Davis JC, Ilegbodu D, Kochis J, Asmar L. Comparison of menopausal symptoms during the first year of adjuvant therapy with either exemestane or tamoxifen in early breast cancer: report of a Tamoxifen Exemestane Adjuvant Multicenter trial substudy. J Clin Oncol. 2007 Oct 20;25(30):4765-71. doi: 10.1200/JCO.2007.10.8274. PMID 17947724
- [Result] Kelley C. Estrogen and its effect on vaginal atrophy in post-menopausal women. Urol Nurs. 2007 Feb;27(1):40-5. PMID 17390926
- [Result] Chin SN, Trinkaus M, Simmons C, Flynn C, Dranitsaris G, Bolivar R, Clemons M. Prevalence and severity of urogenital symptoms in postmenopausal women receiving endocrine therapy for breast cancer. Clin Breast Cancer. 2009 May;9(2):108-17. doi: 10.3816/CBC.2009.n.020. PMID 19433392
- [Result] Sousa MS, Peate M, Jarvis S, Hickey M, Friedlander M. A clinical guide to the management of genitourinary symptoms in breast cancer survivors on endocrine therapy. Ther Adv Med Oncol. 2017 Apr;9(4):269-285. doi: 10.1177/1758834016687260. Epub 2017 Jan 31. PMID 28491147
- [Result] Robinson PJ, Bell RJ, Christakis MK, Ivezic SR, Davis SR. Aromatase Inhibitors Are Associated With Low Sexual Desire Causing Distress and Fecal Incontinence in Women: An Observational Study. J Sex Med. 2017 Dec;14(12):1566-1574. doi: 10.1016/j.jsxm.2017.09.018. Epub 2017 Oct 21. PMID 29066307
- [Result] Wu JM, Vaughan CP, Goode PS, Redden DT, Burgio KL, Richter HE, Markland AD. Prevalence and trends of symptomatic pelvic floor disorders in U.S. women. Obstet Gynecol. 2014 Jan;123(1):141-148. doi: 10.1097/AOG.0000000000000057. PMID 24463674
- [Result] Islam RM, Oldroyd J, Rana J, Romero L, Karim MN. Prevalence of symptomatic pelvic floor disorders in community-dwelling women in low and middle-income countries: a systematic review and meta-analysis. Int Urogynecol J. 2019 Dec;30(12):2001-2011. doi: 10.1007/s00192-019-03992-z. Epub 2019 Jun 4. PMID 31165221
- [Result] Weintraub AY, Glinter H, Marcus-Braun N. Narrative review of the epidemiology, diagnosis and pathophysiology of pelvic organ prolapse. Int Braz J Urol. 2020 Jan-Feb;46(1):5-14. doi: 10.1590/S1677-5538.IBJU.2018.0581. PMID 31851453
- [Result] Ramaseshan AS, Felton J, Roque D, Rao G, Shipper AG, Sanses TVD. Pelvic floor disorders in women with gynecologic malignancies: a systematic review. Int Urogynecol J. 2018 Apr;29(4):459-476. doi: 10.1007/s00192-017-3467-4. Epub 2017 Sep 19. PMID 28929201
- [Result] Rutledge TL, Heckman SR, Qualls C, Muller CY, Rogers RG. Pelvic floor disorders and sexual function in gynecologic cancer survivors: a cohort study. Am J Obstet Gynecol. 2010 Nov;203(5):514.e1-7. doi: 10.1016/j.ajog.2010.08.004. Epub 2010 Sep 24. PMID 20869691
- [Result] Neron M, Bastide S, Tayrac R, Masia F, Ferrer C, Labaki M, Boileau L, Letouzey V, Huberlant S. Impact of gynecologic cancer on pelvic floor disorder symptoms and quality of life: an observational study. Sci Rep. 2019 Feb 19;9(1):2250. doi: 10.1038/s41598-019-38759-5. PMID 30783163
- [Result] Wiegersma M, Panman CM, Berger MY, De Vet HC, Kollen BJ, Dekker JH. Minimal important change in the pelvic floor distress inventory-20 among women opting for conservative prolapse treatment. Am J Obstet Gynecol. 2017 Apr;216(4):397.e1-397.e7. doi: 10.1016/j.ajog.2016.10.010. Epub 2016 Oct 15. PMID 27751796
- [Result] Fallowfield LJ, Bliss JM, Porter LS, Price MH, Snowdon CF, Jones SE, Coombes RC, Hall E. Quality of life in the intergroup exemestane study: a randomized trial of exemestane versus continued tamoxifen after 2 to 3 years of tamoxifen in postmenopausal women with primary breast cancer. J Clin Oncol. 2006 Feb 20;24(6):910-7. doi: 10.1200/JCO.2005.03.3654. PMID 16484701